CLINICAL TRIAL: NCT05018052
Title: Characteristics and Predictors of Early and Late Cardiovascular Complications of Covid-19 Patients - the PoLoCOV-Study (Polish LONG-COVID Cardiovascular Study)
Brief Title: Early and Late Complications of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Michal Chudzik (Other)
Responsible Party: Sponsor-Investigator, Michal Chudzik, Medical Doctor, Cardiologist, Medical Director Ambulatory Clinic, Saint Family Hospital Medical Center
Organization: Saint Family Hospital Medical Center (Other)
Other Study IDs: Stop-Covid/1/2021
Record Dates: First submitted 2021-08-23; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Covid19; LONG-COVID
Keywords: Covid19; Covid complications; Long-Covid; Chronic Fatigue Syndrome
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a serious respiratory disease that results from infection with a newly discovered coronavirus (SARS-COV-2). Unfortunately, COVID-19 is not only a short-term infection. Patients (pts) recovering from SARS-COV2 infection complain of persisting symptoms including: fatigue, diffuse myalgia and weakness, which may lead to chronic fatigue syndrome and as well as many other complications.

The vast majority of COVID-19 patients remaining in isolation/quarantine, due to the mild course of the disease, do not require hospitalization. In this group of patients, the course of COVID-19 is very different - from asymptomatic patients to very severe and long lasting symptoms also with a decrease in saturation.

There are many studies describing the course and complications of patients hospitalized due to COVID-19. There is little published data on how non-hospitalized patients get sick and what are the early and late complications of SARS-CoV-2 infection. In addition, many patients remain ill even many months after COVID-19, entering what is known as LONG-COVID.

Therefore, the STOP-COVID Registry was established. The purpose of the Registry is to assess the course of COVID-19 infection, early and late cardiovascular complications of COVID-19 in patients with and without hospitalization. In addition, the purpose of the STOP-COVID Registry is to assess the incidence of LONG-COVID with all other complications and to identify predictive factors.

DETAILED DESCRIPTION:
The following patients are included in the Registry: Patients 18 years and older diagnosed with COVID-19, in accordance with the current guidelines of the Ministry of Health of Poland, after full recovery (resolution of clinical symptoms, minimum 14 days after last symptoms). The Registry includes patients with and without hospitalization .

Approval from the Bioethics Committee of Lodz Regional Medical Chamber to conduct the Registry was obtained.

The Registry was held at the: Saint Family Hospital Medical Center, Lodz, Poland Patient information, course of the disease, post-COVID-19 complaints, comorbidities and current treatment were collected at visit "0" within 4-8 weeks after the end of COVID-19.

Subsequently, patients were ordered the following tests:

* 12-lead ECG
* 24-hour Holter ECG monitoring
* 24-hour Holter blood pressure monitoring
* Echocardiographic of the Heart assessment
* Biochemical tests: Lipid Profile (total cholesterol, LDL fraction, HDL, triglycerides), glucose or glycosylated hemoglobin (HbA1c) level, D-dimers.

In patients with indications, the following were additionally performed: MRI of the heart, Angio CT of pulmonary vessels, Angio CT of coronary vessels or other diagnostic tests. Depending on the indications of the pts, they were referred for other tests and specialist consultations. All pts were diagnosed and treated in accordance with the current recommendations of the European Cardiology Society (ESC) and Polish Cardiac Society (PCS).

If any abnormalities were found, patients were treated in accordance with the current ESC guidelines. In the event of complications after COVID-19, each patient will be treated in accordance with current guidelines and recommendations, in accordance with current medical knowledge.

After a period of 3 months after COVID-19, new symptoms that appeared after COVID-19, remained and/or worsened after COVID-19 were assessed at the follow-up visit, based on the patient's interview. If such symptoms occurred, patients were classified as LONG-COVID. Symptoms that may have resulted from the severity of the underlying condition were not classified as LONG-COVID.

Patients with LONG-COVID, after excluding complications/contraindications, will be referred to the post-COVID rehabilitation program. This program covers a comprehensive range of rehabilitation with dietary and psychological consultations. Patients referred to the rehabilitation program will constitute the REHA-STOP-COVID group. The rehabilitation program will last 6 weeks. At the beginning and at the end of the program, each patient will have fitness assessment performed with the following tests:

* oxygen saturation assessment performed with a pulse oximeter;
* physical capacity assessment with 6 minute walking test (6MWT)
* Dyspnea assessment with modified 0-10 Borg scale
* Fatigue assessment with Modified Fatigue Impact Scale (MFIS)
* Muscle Strength Assessment
* lower extremity function and mobility with Short Physical Performance Battery test (SPPB)

Annual reassessment of all patients is planned for 5 years after COVID-19.

During the control visits, patients will be ordered the following:

* Clinical evaluation with health assessment, comorbidities and symptoms that may be due to a history of COVID-19
* 12-lead ECG
* 24-hour Holter ECG monitoring
* 24-hour Holter blood pressure monitoring
* Echocardiographic of the Heart assessment
* Biochemical tests: Lipid Profile (total cholesterol, LDL fraction, HDL, triglycerides), glucose or glycosylated hemoglobin (HbA1c).

Additionally, a questionnaire will be completed by the patient with an assessment of his/her health, weight, height, BMI, risk factors for cardiovascular diseases (smoking, alcohol abuse), physical activity, all medications that the patient takes, whether the patient was re-infected with SARS-CoV in the past years (date) , whether the patient was vaccinated (with full vaccination date).

Each patient from the STOP-COVID program, in the event of deterioration of health and / or the appearance of new ailments, may be referred for the consultation to the Saint Family Hospital Medical Center by a GP and/or another specialist during the whole period of the study.

During the entire study period, the following will be registered in the medical database:

1. Any new medical event assessed by 2 doctors as a complication after COVID-19
2. Any hospitalization related to complications of COVID-19 as well as any other reason
3. Each severity has already been diseases diagnosed and treated, with information whether it required correction / modification of the current treatment
4. Any newly diagnosed diseases
5. Any abnormalities in the results of diagnostic examinations, laboratory tests and consultations

ELIGIBILITY:
Inclusion Criteria:

Patients after COVID-19, 18 years and older

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and older diagnosed with COVID-19, after full recovery (resolution of clinical symptoms, minimum 14 days after last symptoms), with and without hospitalization .
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Early and Late COVID-19 cardio-vascular complications | 5 years
  Early and Late COVID-19 cardio-vascular complications
Predictors of Long-Covid Cardio-Vascular complications | 5 years
  Predictors of Long-Covid Cardio-Vascular complications
SCORE - algorithm to help to predict the highest risk of Long-Covid complications | 5 years
  SCORE - algorithm to help to predict the highest risk of Long-Covid complications

SECONDARY OUTCOMES:
Detailed patients' characteristics and differences in those with and without Long-Covid complications | 5 years
  Detailed patients' characteristics and differences in those with and without Long-Covid
Definition and characteristics of the early and Late COVID-19 complications | 5 years
  Definition and characteristics of the early and Late COVID-19 complications
Comparison of complications and Long-Covid depending on the severity of the course of COVID-19 COVID-19, comorbidities | 5 years
  Comparison of complications and Long-Covid depending on the severity of the course of COVID

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center, Saint Family Hospital, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Babicki M, Kapusta J, Kolat D, Kaluzinska-Kolat Z, Mastalerz-Migas A, Jankowski P, Chudzik M. Cardiac symptoms in patients 3-6 months after contracting COVID-19- data from the polish STOP-COVID registry. BMC Infect Dis. 2025 Apr 9;25(1):489. doi: 10.1186/s12879-025-10774-0. PMID 40205590
- [Derived] Kapusta J, Chudzik M, Kaluzinska-Kolat Z, Kolat D, Burzynska M, Jankowski P, Babicki M. Do selected lifestyle parameters affect the severity and symptoms of COVID-19 among elderly patients? The retrospective evaluation of individuals from the STOP-COVID registry of the PoLoCOV study. J Infect Public Health. 2023 Jan;16(1):143-153. doi: 10.1016/j.jiph.2022.12.008. Epub 2022 Dec 12. PMID 36521330
- See also: Related Info — http://www.stop-covid.pl